CLINICAL TRIAL: NCT06182670
Title: The Role of a New Prosthodontics Device in Hard and Soft Tissue Changes After Subcrestal Implant Placement: 12-months, Parallel, Randomized Clinical Trial
Brief Title: The Role of a New Prosthodontics Device in Hard and Soft Tissue Changes After Subcrestal Implant Placement
Acronym: NABUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Magda Mensi, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NABUT NP 4078
Record Dates: First submitted 2023-12-10; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Oral Implants; Abutment; Subcrestal

STUDY DESIGN:
Intervention Model Description: Monocentric, single blinded, randomized clinical trial, parallel design.
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcrestal implant and gingival former abutment (GFA) (Experimental): The subjects receive a subcrestal implant and a prosthodontic device (GFA) immediately during the surgery. The GFA will not be removed upon prosthetic load. It will be an integral part of the prosthetic finalization.
  Interventions: Device: Gingival Former Abutment; Procedure: Subcrestal Implant; Device: Prosthetic Crown
- Crestal implant and traditional abutment (Active Comparator): The subjects receive a crestal implant and healing abutment. The healing abutment will be replaced by a definitive abutment to the prosthetic load.
  Interventions: Device: Healing Abutment; Device: Prosthetic Crown; Procedure: Crestal Implant

INTERVENTIONS:
Device: Gingival Former Abutment — GFA is positioned on the sub-crestal implant during the surgery and it is no longer removed. This follows the "one abutment one time" concept and should prevent bone loss and transmucosal tunnel.
  Arms: Subcrestal implant and gingival former abutment (GFA)
Procedure: Subcrestal Implant — Placement of the endosseous sub-crestal dental implant through dedicated drills with 35 Newton insertion torque. It is positioned 2 mm under the crestal bone.
  Arms: Subcrestal implant and gingival former abutment (GFA)
Device: Healing Abutment — A healing abutment is positioned on crestal implant during surgery. It is removed at prosthetic finalization.
  Arms: Crestal implant and traditional abutment
Device: Prosthetic Crown — A zirconia prosthetic crown finalizes the implant rehabilitation.
Procedure: Crestal Implant — Placement of the endosseous crestal implant through dedicated drills with 35 Newton insertion torque at level of the alveolar bone.
  Arms: Crestal implant and traditional abutment

SUMMARY:
The present randomized controlled trial aims to assess the influence of a new prosthodontics device (Gingival Former Abutment -GFA) on peri-implant bone loss and soft tissue changes and health after subcrestal oral implant placement.

The participants will be divided in two groups and receive either crestal implant placement and traditional healing abutment or subcrestal implant placement and GFA.

Clinical and radiographic examination will be performed at implant placement surgery, prosthetic load, 6 and 12 months follow-up.

DETAILED DESCRIPTION:
According to current literature, physiological bone loss around oral implants is expected after placement and load (1 mm during the first year and 0.2 mm each subsequent year). Different implant designs and surgical protocols have been tested to minimize bone resorption, and subcrestal implant placement partially seems to overcome this issue. However, if this procedure increases the length of the transmucosal tunnel, increasing the risk of peri-implant soft tissue infection.

The GFA was created to limit both the loss of peri-implant crestal bone and the extension of the transmucosal tunnel. The GFA follows the "one abutment one time" concept, which is believed to limit disturbances of the peri-implant hard and soft tissues healing due to the removal of the traditional healing abutments during prosthetic load procedures. Our objective is to validate or deny this claim.

The study is a monocentric, pragmatic, single-blinded, randomized clinical trial (RCT) of parallel design. The trial will have a one-year duration, with data collection at the surgical phase, at implant load and 6 and 12 months after load. The primary outcome will be radiographical MBL (marginal bone level) changes around the implant. Secondary outcomes will be the assessment of the peri-implant soft tissues.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and sign informed consent.
* Male and female subjects, aged 18-75 years, inclusive.
* Good general health (free of systemic diseases such as diabetes, HIV infection or genetic disorder, ongoing malignant disease of any type that could influence the outcome of the treatment and might interfere with the evaluation of the study objectives).
* Good oral health (no decay, periapical or periodontal lesions, PI and BOP <25%).
* Patient with posterior single missing tooth:

  * for at least 5 months,
  * mandibular or maxillary,
  * intercalated (distance between teeth more than 7.5 mm),
  * at least 11 mm of height residual bone (from bone crest to maxillary sinus or inferior alveolar nerve),
  * at least 5 mm of bone width (buccal - palatal/lingual).
* Availability for the 12-month duration of the study.

Exclusion Criteria:

* Not willing to follow the agreed protocol.
* Presence of orthodontic appliances.
* Smokers more than 10 cigarettes per day.
* Chronic obstructive pulmonary disease and asthma.
* Tumors or significant pathology of the soft or hard tissues of the oral cavity.
* Current radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Parafunctions like bruxism.
* Previous interventions to increase bone thickness in the implant area.
* Current or past assumption of medications that may influence surgical therapy and/or interfere with healing following surgical treatment.
* Systemic diseases that constitute a contraindication to surgical therapy and/or interfere with healing following surgical treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Change in Marginal Bone Level (MBL) | Surgery, 3, 9 and 15 months
  The reabsorption of the bone measured through radiographically change on standardised radiographs. Baseline values will be compared to the values recorded in the follow-up visits.

SECONDARY OUTCOMES:
Change in PD (periodontal depth) (implant site) | 3, 9 and 15 months
  Change in periodontal depth value (from the gingival margin to the bottom of the pocket). Baseline values will be compared to the values recorded in the follow-up visits.
Change in REC (Clinical Gingival Recession) (implant site) | 3, 9 and 15 months
  Change in recession value should be calculated. Baseline values will be compared to the values recorded in the follow-up visits.
Change in BOP (Bleeding on Probing) (implant site) | 3, 9 and 15 months
  Change in percentage of sites positive to bleeding on probing (4 point each situ). Baseline values will be compared to the values recorded in the follow-up visits.
Change in PI (Plaque Index) (implant site) | 3, 9 and 15 months
  Change in percentage of site with plaque (4 point each situ). Baseline values will be compared to the values recorded in the follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Mensi, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Magda Mensi, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT06182670/Prot_SAP_000.pdf